CLINICAL TRIAL: NCT06282809
Title: The HistoSonics Edison™ System for Treatment of Pancreatic Adenocarcinoma Using Histotripsy
Acronym: GANNON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HistoSonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP3325
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Pancreas Cancer; Adenocarcinoma of the Pancreas; Pancreatic Cancer; Tumor of Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective multi-center, single-arm, feasibility trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- HistoSonics System (Experimental)
  Interventions: Device: HistoSonics Edison™ System for the treatment of pancreatic adenocarcinoma using histotripsy

INTERVENTIONS:
Device: HistoSonics Edison™ System for the treatment of pancreatic adenocarcinoma using histotripsy — Histotripsy is a non-thermal, mechanical process of focused ultrasound used to mechanically destroy targeted soft tissue.

SUMMARY:
The purpose of this trial is to evaluate the safety of the HistoSonics Edison System for the destruction of pancreatic adenocarcinomas using histotripsy.

DETAILED DESCRIPTION:
This is a prospective multi-center, single-arm, feasibility trial designed to evaluate the safety of the HistoSonics Edison System for the destruction of pancreatic adenocarcinoma tumors in patients who are diagnosed with unresectable locally advanced (Stage 3) or oligometastatic disease (Stage 4).

The type of design is exploratory and is considered interventional. Following histotripsy, subjects will undergo imaging ≤36-hours post-index procedure. Additionally, subjects will be followed at 7-day, 14-day, 30-day, 60-day, 120-day, and 180-day timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age.
2. Subject has signed the Ethics Committee (EC) approved trial Informed Consent Form (ICF) prior to any trial related tests/procedures and is willing to comply with trial procedures and required follow-up assessments.
3. Subject is diagnosed with unresectable pancreatic adenocarcinoma (locally advanced [Stage 3] or oligometastatic disease [Stage 4]) confirmed via CT or MR imaging ≤14 days prior to the planned index procedure.

   NOTE: If Stage 4 disease, there must be ≤5 metastatic tumors, the tumors must be located only in the liver and/or lung, and the metastatic tumors must be stable.
4. Subject is not a surgical candidate and has received chemotherapy ≥8 weeks.
5. Subject can tolerate general anesthesia.
6. Subject has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) grade 0-1 at baseline.
7. Subject meets the following criteria ≤14 days prior to the planned index procedure date:

   * Hemoglobin ≥ 9 g/dL,
   * Neutrophil count >1.0 x 10^9/L,
   * Platelet >50 x 10^9/L,
   * Total bilirubin ≤2.5x Institutional Upper Limit of Normal (IULN),
   * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.5x IULN,
   * International Normalized Ratio (INR) value <1.5,
   * Serum creatinine <2.0mg/dL or an estimated glomerular filtration rate (eGFR) ≥45mL/min.
8. The targeted pancreatic tumor is ≥2 cm in longest diameter.
9. The planned histotripsy treatment volume is ≥1.0 cm from any portion of the duodenum, small intestine, stomach, or colon as visualized on ultrasound, and CT, or MR imaging.
10. Subject has an adequate acoustic window to visualize targeted tumor using the HistoSonics Edison System.
11. Subject will undergo histotripsy treatment of only one (1) tumor during the index procedure, regardless of how many tumors are present in the pancreas.

Exclusion Criteria:

1. Subject is pregnant or planning to become pregnant or nursing (lactating) during the trial period.
2. Subject has had prior pancreatic, bilioenteric, or gastric surgery.
3. Subject is being actively treated in another pharmaceutical or device trial that has not completed its primary endpoint prior to the index procedure or may interfere with the primary outcome measure of this trial.
4. Subject has an uncorrectable coagulopathy.
5. Subject has a life expectancy of less than six (6) months.
6. Subject has a biliary or pancreatic stent and/or percutaneous biliary tube that encompasses the planned histotripsy treatment volume.
7. Subject has metastases to organs other than the liver and/or lung (e.g., bone, brain, peritoneum).
8. Subject has a known sensitivity to contrast media and cannot be adequately pre-medicated.
9. Subject has an active duodenal or gastric ulcer requiring medical management.
10. Subject is undergoing active chemotherapy for any cancer ≤7 days prior to planned index procedure date.*
11. Subject is undergoing active immunotherapy or targeted therapies ≤30 days prior to planned index procedure date.
12. Subject's targeted tumor has had prior locoregional therapy (e.g., ablation, embolization, or radiation).
13. Subject has a planned cancer treatment (e.g., pancreatic surgery, targeted therapy, immunotherapy) exclusive of chemotherapy, ≤30 days post index procedure.
14. Subject has planned chemotherapy ≤14 days post index procedure.*
15. Subject has not recovered (CTCAE grade 2 or better) from chemotherapy or immunotherapy related toxicities (exclusive of alopecia, neuropathy, and exocrine insufficiency).
16. In the investigator's opinion, histotripsy is not a treatment option for the subject.
17. Subject has a concurrent condition that could jeopardize the safety of the subject or compliance with the protocol.
18. Subject's tumor is not treatable by the System's working ranges (refer to User Guide).

(*) Subject must not be off chemotherapy >21 days in total.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of the HistoSonics Edison System for the destruction of pancreatic adenocarcinomas using histotripsy | 30 days post histotripsy procedure
  Index procedure-related complications ≤30 days post index procedure, graded using Clavien-Dindo Classification and Common Terminology Criteria for Adverse Events (CTCAE). [Clinical Events Committee Adjudicated]

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No